CLINICAL TRIAL: NCT03529630
Title: Breastfeeding Success With the Use of the WHO Syringe Technique for Management of Inverted Nipples in Lactating Women: a Study Protocol for a Randomized Controlled Trial
Brief Title: Breastfeeding Success With the Use of the WHO Syringe Technique for Management of Inverted Nipples in Lactating Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Mona Nabulsi, Professor of Clinical Pediatrics, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED.MN.15
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Breastfeeding; Inverted Nipple
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inverted syringe (Experimental): Participants in this arm will use of the inverted syringe before each breastfeeding starting from the first feed after delivery and continued as long as needed by the mother.
  Interventions: Other: Inverted syringe
- Standard of care (No Intervention): Participants in the control group will receive standard medical care as dictated by their obstetricians. Any advice regarding infant nutrition or treatment of inverted nipples will be left to the primary physician, including possible use of the inverted syringe technique. .

INTERVENTIONS:
Other: Inverted syringe — Application of mild suction over the mother's inverted nipple using an inverted syringe before each breastfeeding.
  Arms: Inverted syringe

SUMMARY:
Breastfeeding is the ideal infant nutrition recommended by governmental and medical professional organizations. Yet, women with inverted nipples often face difficulties in breastfeeding that ultimately force them to prematurely terminate breastfeeding. This open-label randomized clinical trial aims to investigate the effectiveness of the use of the inverted syringe technique on exclusive breastfeeding success in women with inverted nipples, as compared to standard of care.

DETAILED DESCRIPTION:
Breastfeeding is the ideal infant nutrition recommended by governmental and medical professional organizations. Its benefits to infants and their mothers are many including protection from infections, certain malignancies and chronic diseases, as well as improved growth, development, cognition and intelligence for children. Yet, women with inverted nipples often face difficulties in breastfeeding that ultimately force them to prematurely terminate breastfeeding. The main treatment of severely inverted nipples is surgical sectioning of the lactiferous ducts at the expense of breast's function. Several conservative measures have also been used for the less severe (grades 1 and 2) inverted nipples such as application of Hoffman Exercises and Woolwich Breast Shields, which have failed to prove their worth. The modified syringe technique is a conservative means for the correction of inverted nipples that was reported in a single case series of 8 women, with high success rates in infant latching (7/8) and exclusive breastfeeding (6/8). It is a simple, inexpensive, portable, safe, and easily learned method that can be performed by mothers as often as required.

This open-label randomized clinical trial aims to investigate the effectiveness of the use of inverted syringe on the 1-month exclusive breastfeeding rate in women with inverted nipples. We hypothesize that in women with grades 1 and 2 inverted nipples, the use of the modified syringe technique soon after delivery, as opposed to the standard of care, will significantly improve breastfeeding rates at 1 month postpartum. We will recruit 100 healthy women at ≥37 weeks of gestation with grades 1 or 2 inverted nipples from the Women's Health Center and the obstetrics outpatient department at AUBMC. They will be randomly allocated to a control group (standard of care) or to the intervention group (inverted syringe). Data will be collected at baseline (socio-demographic variables, inverted nipple grading) and at 1, 3, and 7 days postpartum about infant feeding method, and adverse events. Mothers will be contacted at 1, 3 and 6 months regarding infant feeding method, maternal satisfaction, infant's weight gain and adverse events. The association between breastfeeding success at 1 month and the use of the inverted syringe will be investigated using multivariate regression models. Findings from this study, if positive, will provide much needed evidence for a safe, affordable, readily available and simple intervention to treat inverted nipples and improve breastfeeding practice among affected women.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women in their 37th week of gestation or more with grade 1 or 2 inverted nipples
2. Able to read and write
3. Singleton or twin pregnancy An inverted nipple is defined as a condition in which the nipple is pulled inward into the breast instead of pointing outward, classified according to Han and Hong [11].

Exclusion Criteria:

1. Women with grade 3 inverted nipples
2. Previous breast surgery affecting the breast anatomy
3. High risk pregnancies
4. Medical conditions that could interfere with breastfeeding such as critical maternal condition
5. Newborns with congenital malformations that may interfere with breastfeeding such as esophageal atresia, cleft lip &/or palate
6. Women choosing artificial milk as their preferred infant nutrition.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
One month exclusive breastfeeding rate | 1 month postpartum
  Proportion of mothers who are exclusively breastfeeding

SECONDARY OUTCOMES:
3-month exclusive breastfeeding rate | 3 months postpartum
  Proportion of mothers who are exclusively breastfeeding
6-month exclusive breastfeeding rate | 6 months postpartum
  Proportion of mothers who are exclusively breastfeeding
Nipple eversion rate | 1 month postpartum
  Proportion of mothers with everted nipples
Successful latching | 1 month postpartum
  Proportion of infants with successful latching while breastfeeding
1-month mixed feeding rate | 1 month postpartum
  Proportion of infants on mixed feeding
3-month mixed feeding rate | 3 months postpartum
  Proportion of infants on mixed feeding
6-month mixed feeding rate | 6 months postpartum
  Proportion of infants on mixed feeding
Breastfeeding-associated complications | 1 week postpartum
  Rate of breastfeeding-associated complications such as sore nipple, mastitis, pain, bleeding, breast engorgement
Breastfeeding-associated complications | 1 month postpartum
  Rate of breastfeeding-associated complications such as sore nipple, mastitis, pain, bleeding, breast engorgement
Breastfeeding-associated complications | 3 months postpartum
  Rate of breastfeeding-associated complications such as sore nipple, mastitis, pain, bleeding, breast engorgement
Breastfeeding-associated complications | 6 months postpartum
  Rate of breastfeeding-associated complications such as sore nipple, mastitis, pain, bleeding, breast engorgement
Maternal satisfaction with breastfeeding | 1 week postpartum
  Maternal satisfaction with breastfeeding assessed with the validated Maternal Breastfeeding Evaluation Scale (MBFES). The scale measures the overall maternal perceived quality with the breastfeeding experience. The scale has a Cronbach's alpha of 0.93. It is composed of 3 subscales: maternal enjoyment/role attainment, infant satisfaction/growth and lifestyle/body image. The corresponding Cronbach's alphas of the subscales are 0.93, 0.88 and 0.80 respectively. The overall score may range from 30 (least satisfied) to 150 (most satisfied).
Maternal quality of life | 1 month postpartum
  Maternal quality of life assessed with the validated Postpartum Quality of Life instrument

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Sharing of anonymized IPD is possible upon request from the principal investigator after 1 year from publication of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After December 2021.
Access Criteria: Request data sharing from the principal investigator.

REFERENCES:
- [Background] Binns C, Lee M, Low WY. The Long-Term Public Health Benefits of Breastfeeding. Asia Pac J Public Health. 2016 Jan;28(1):7-14. doi: 10.1177/1010539515624964. PMID 26792873
- [Background] Victora CG, Horta BL, Loret de Mola C, Quevedo L, Pinheiro RT, Gigante DP, Goncalves H, Barros FC. Association between breastfeeding and intelligence, educational attainment, and income at 30 years of age: a prospective birth cohort study from Brazil. Lancet Glob Health. 2015 Apr;3(4):e199-205. doi: 10.1016/S2214-109X(15)70002-1. PMID 25794674
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Yan J, Liu L, Zhu Y, Huang G, Wang PP. The association between breastfeeding and childhood obesity: a meta-analysis. BMC Public Health. 2014 Dec 13;14:1267. doi: 10.1186/1471-2458-14-1267. PMID 25495402
- [Background] Belfort MB, Rifas-Shiman SL, Kleinman KP, Guthrie LB, Bellinger DC, Taveras EM, Gillman MW, Oken E. Infant feeding and childhood cognition at ages 3 and 7 years: Effects of breastfeeding duration and exclusivity. JAMA Pediatr. 2013 Sep;167(9):836-44. doi: 10.1001/jamapediatrics.2013.455. PMID 23896931
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Kramer MS, Kakuma R. Optimal duration of exclusive breastfeeding. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD003517. doi: 10.1002/14651858.CD003517.pub2. PMID 22895934
- [Background] SKOOG T. An operation for inverted nipples. Br J Plast Surg. 1952 Apr;5(1):65-9. doi: 10.1016/s0007-1226(52)80008-6. No abstract available. PMID 14944774
- [Background] Terrill PJ, Stapleton MJ. The inverted nipple: to cut the ducts or not? Br J Plast Surg. 1991 Jul;44(5):372-7. doi: 10.1016/0007-1226(91)90152-a. PMID 1873618
- [Background] Han S, Hong YG. The inverted nipple: its grading and surgical correction. Plast Reconstr Surg. 1999 Aug;104(2):389-95; discussion 396-7. doi: 10.1097/00006534-199908000-00010. PMID 10654681
- [Background] Alexander JM, Grant AM, Campbell MJ. Randomised controlled trial of breast shells and Hoffman's exercises for inverted and non-protractile nipples. BMJ. 1992 Apr 18;304(6833):1030-2. doi: 10.1136/bmj.304.6833.1030. PMID 1586788
- [Background] McGeorge DD. The "Niplette": an instrument for the non-surgical correction of inverted nipples. Br J Plast Surg. 1994 Jan;47(1):46-9. doi: 10.1016/0007-1226(94)90117-1. PMID 8124566
- [Background] Chakrabarti K, Basu S. Management of flat or inverted nipples with simple rubber bands. Breastfeed Med. 2011 Aug;6(4):215-9. doi: 10.1089/bfm.2010.0028. Epub 2011 Jan 8. PMID 21214390
- [Background] Kesaree N, Banapurmath CR, Banapurmath S, Shamanur K. Treatment of inverted nipples using a disposable syringe. J Hum Lact. 1993 Mar;9(1):27-9. doi: 10.1177/089033449300900127. PMID 8489719
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Leff EW, Jefferis SC, Gagne MP. The development of the Maternal Breastfeeding Evaluation Scale. J Hum Lact. 1994 Jun;10(2):105-11. doi: 10.1177/089033449401000217. PMID 7619250
- [Background] Riordan JM, Woodley G, Heaton K. Testing validity and reliability of an instrument which measures maternal evaluation of breastfeeding. J Hum Lact. 1994 Dec;10(4):231-5. doi: 10.1177/089033449401000416. PMID 7619277
- [Background] Hill PD, Aldag JC, Hekel B, Riner G, Bloomfield P. Maternal Postpartum Quality of Life Questionnaire. J Nurs Meas. 2006 Winter;14(3):205-20. doi: 10.1891/jnm-v14i3a005. PMID 17278340
- [Background] Nabulsi M, Hamadeh H, Tamim H, Kabakian T, Charafeddine L, Yehya N, Sinno D, Sidani S. A complex breastfeeding promotion and support intervention in a developing country: study protocol for a randomized clinical trial. BMC Public Health. 2014 Jan 15;14:36. doi: 10.1186/1471-2458-14-36. PMID 24428951
- [Derived] Nabulsi M, Ghanem R, Smaili H, Khalil A. The inverted syringe technique for management of inverted nipples in breastfeeding women: a pilot randomized controlled trial. Int Breastfeed J. 2022 Feb 5;17(1):9. doi: 10.1186/s13006-022-00452-1. PMID 35123525
- [Derived] Nabulsi M, Ghanem R, Abou-Jaoude M, Khalil A. Breastfeeding success with the use of the inverted syringe technique for management of inverted nipples in lactating women: a study protocol for a randomized controlled trial. Trials. 2019 Dec 16;20(1):737. doi: 10.1186/s13063-019-3880-8. PMID 31842992